CLINICAL TRIAL: NCT05748197
Title: A Phase I Study of ADCLEC.syn1 CAR T Cells in Adult Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: A Study of ADCLEC.syn1 in People With Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-002
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Relapsed; Refractory; ADCLEC.syn1 CAR T cells; Cyclophosphamide; Fludarabine; 23-002
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Intervention Model Description: This is a phase I, open-label, dose-escalation/dose expansion trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADCLEC.syn1 CAR T cells (Experimental): The dose escalation cohort size of 3 patients in each cohort will be infused with escalating doses of ADCLEC.syn1 CAR T cells to inform the RP2D. There are 4 planned flat-dose levels: 25 × 10^6, 75 × 10^6 , 225 × 10^6 , and 450 × 10^6 CAR T cells and 1 de-escalation dose: 10 × 10^6 CAR T cells. After dose escalation, one or two dose levels will be selected for dose expansion cohort(s).Two to 7 days following completion of the conditioning chemotherapy, the frozen CAR T cells will be thawed and administered. Conditioning chemotherapy may occur either outpatient or inpatient, and T cell infusions will occur as inpatient. Up to approximately 12 additional patients each if two doses are selected or approximately 16 additional patients, if one dose is selected, will be treated in the dose expansion phase to determine RP2D.
  Interventions: Biological: ADCLEC.syn1 CAR T cells; Drug: Conditioning chemotherapy

INTERVENTIONS:
Biological: ADCLEC.syn1 CAR T cells — There are 4 planned flat-dose levels: 25 × 10^6, 75 × 10^6 , 225 × 10^6 , and 450 × 10^6 CAR T cells and 1 de-escalation dose: 10 × 10^6 CAR T cells.
Drug: Conditioning chemotherapy — Fludarabine 30 mg/m2 daily for 3 days and cyclophosphamide 500 mg/m2 daily for 3 days.

SUMMARY:
The purpose of this study is to test the safety of ADCLEC.syn1 CAR T cells in people with relapsed or refractory AML. The researchers will try to find the highest dose of ADCLEC.syn1 CAR T cells that causes few or mild side effects in participants. Once the researchers find this dose, it will test it in a new group of participants to see if it is effective in treating their relapsed/refractory AML.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age at the time of signing informed consent.
2. Patients must have R/R AML. The following disease status will be eligible for the study:

   a. Refractory AML is defined as failure to achieve a CR, CRh or CRi after one of the following regimens: i. At least one course of standard intensive induction chemotherapy (e.g., 7+3, MEC, HiDAC, etc.) or hypomethylating agent (HMA) or low dose cytarabine-based combination regimen including but not limited to venetoclax (e.g. venetoclax in combination with azacytidine, decitabine or cytarabine) ii. Four cycles of HMA monotherapy b. Relapsed AML is defined the appearance of ≥5% blasts in the bone marrow or peripheral blood at any time after achieving a CR, CRh, or CRi.
3. ECOG performance status 0 or 1.
4. Subjects must have a suitable stem cell donor identified who may donate cells in the event that the subject needs to undergo an allogeneic HSCT for rescue from prolonged marrow aplasia.

   Donor may be from related or unrelated matched source, haplo or cord, and must be found to be suitable according to the institution's standard criteria.
5. Adequate organ function defined as:

   1. Serum creatinine <2.0 mg/100 mL.
   2. Total bilirubin <2.0 mg/100 mL, unless benign congenital hyperbilirubinemia or due to leukemia organ involvement
   3. AST and/or ALT ≤5 × ULN, unless considered due to leukemic organ involvement.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia.
2. Radiologically-detected or symptomatic CNS disease or CNS 3 disease (i.e., presence of ≥5/µL WBCs in CSF). Subjects with adequately treated CNS leukemia are eligible.
3. Oxygen saturation <90% on room air.
4. Patients with prior allogeneic HSCT are allowed as long as HSCT occurred > 3 months of signing ICF and without ongoing requirement for systemic graft-versus-host therapy.
5. Treatment with clofarabine or cladribine within 3 months prior to leukapheresis
6. The following medications are excluded:

   1. Steroids: Therapeutic doses of corticosteroids (greater than 10mg daily of prednisone or its equivalent) within 7 days of leukapheresis or 72 hours prior to CAR T cell infusion.
   2. Chemotherapy: Bridging chemotherapy including venetoclax must be discontinued at least 1 week prior to administration of conditioning chemotherapy, but FDA-approved oral targeted therapies such as IDH1/2, FLT3, and menin inhibitiors as well as hydroxyurea can be continued until at least 24 hours prior to the start of conditioning chemotherapy
7. Clinically significant cardiovascular disease, including stroke or myocardial infarction within 6 months prior to first study medication; or the presence of unstable angina or congestive heart failure of New York Heart Association Grade 2 or higher; or cardiac ejection fraction <40%.
8. Uncontrolled clinically significant infections such as ongoing fever for 48 hours, persistent bacteremia or requiring new supplemental oxygen.
9. Positive serologic test results for HIV.
10. Acute or chronic HBV infection as assessed by serologic (HBVsAg) or PCR results, defined as HBVsAg+, HBVcAb+, HBV PCR+.
11. Acute or chronic HCV infection as assessed by serologic (HCV ab) or PCR results, defined as HCV Ab+ with reflex to positive HCV PCR.
12. Active second malignancy that requires systemic treatments, with the exception of malignancy treated with curative intent and without evidence of disease for >2 years before screening.
13. Live vaccine within 4 weeks prior to leukapheresis
14. Pregnant or lactating/breastfeeding women
15. Any prior or ongoing condition/issue that in the opinion of the investigator would make the patient ineligible for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2028-04-18 (Estimated); Study Completion 2028-04-18 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 2 years
  Dose escalation of ADCLEC.syn1 CAR T cells will follow Bayesian optimal interval (BOIN) design to inform dose-escalation decisions and potential maximum tolerated dose (MTD) estimation. Patients will be enrolled in cohorts of 3.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Commack - Suffolk (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Background] Haubner S, Mansilla-Soto J, Nataraj S, Kogel F, Chang Q, de Stanchina E, Lopez M, Ng MR, Fraser K, Subklewe M, Park JH, Wang X, Riviere I, Sadelain M. Cooperative CAR targeting to selectively eliminate AML and minimize escape. Cancer Cell. 2023 Nov 13;41(11):1871-1891.e6. doi: 10.1016/j.ccell.2023.09.010. Epub 2023 Oct 5. PMID 37802054
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm